CLINICAL TRIAL: NCT06566118
Title: Effects of Transcutaneous Vagus Nerve Stimulation on Recovery After Sports Activity in Young Athletes
Brief Title: Effects of Transcutaneous Vagus Nerve Stimulation on Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Ali Karaağaç, Principal Investigator, Istanbul Gelisim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IGU-FTR-AK-01
Record Dates: First submitted 2024-08-15; First posted 2024-08-22 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Fatigue; Recovery, Psychological
Keywords: Auricular Vagus Nerve Stimulation; Athlete; Recovery
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Uncontrolled study with the same sample in two groups
Who Masked: Participant
Masking Description: During the application to the group that would receive sham auricular vagus nerve stimulation, the device was shown to the participants while it was being operated, but no current was given to the participants because headphones without conductive properties were used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Active auricular VSS was applied to the participants in Group 1 after exercise loading.
  Interventions: Device: Auricular Vagus Nerve Stimülation
- Sham Group (Sham Comparator): Sham auricular VSS was applied to the participants in Group 2. During the application, the device was shown to the participants while it was being operated, but no current was given to the participants because non-conductive headphones were used.
  Interventions: Device: Sham Auricular Vagus Nerve Stimülation

INTERVENTIONS:
Device: Auricular Vagus Nerve Stimülation — After exercise loading, active ear VSS was applied to Group 1. Application was made simultaneously in both ears, with a 300 microsecond pulse duration, a biphasic asymmetric waveform, and a frequency of 25 Hz, for a total of 20 minutes. All assessments were recorded 3 times: at the beginning of the test, after exercise loading, and after active VSS application.
  Arms: Intervention Group
Device: Sham Auricular Vagus Nerve Stimülation — After the exercise challenge, Group 2 underwent sham VSS. Device parameters were set to the same as Group 1 (300 microsecond pulse duration, biphasic asymmetric waveform, and 25 Hz frequency). Both headphones were worn for a total of 20 minutes. However, the participant heard only the device's power-on tone and received no current. All assessments were recorded three times: at the beginning of the test, after the exercise challenge, and after sham VSS.
  Arms: Sham Group

SUMMARY:
During the recovery process, the activity of the sympathetic system decreases, while the activity of the parasympathetic system increases. In line with this information, the nervous system can be regulated in a noninvasive and practical way by using transcutaneous auricular vagus nerve stimulation in order to achieve rapid recovery in the athlete after the activity.

DETAILED DESCRIPTION:
In sports where physical loads are high, athletes can usually participate in more than one training or race during the day. Such work increases the athlete's fatigue, affects their performance and can cause serious declines. Therefore, an efficient and effective recovery process after high-intensity work and training that causes a decrease in performance is also very important for the athlete's next performance.

With the start of sports activity or exercise, sympathetic activation in the body increases and after a while reaches a plateau value at maximum activity. With the end of exercise, this time the suppressed parasympathetic activity begins to increase and the sympathetic system returns to a resting state over time.

There are insufficient studies in the literature investigating the use of Transcutaneous Auricular Vagus Nerve Stimulation on the athletic population. Although it is clear that the application has effects on the sympathetic and parasympathetic nervous systems, more clinical research is needed on athletes. In this study, we aimed to investigate the effects of auricular vagus nerve stimulation (VNS) on vagal activity by examining the effect of transcutaneous auricular vagus nerve stimulation on recovery in amateur athletes through applications such as pulse and SpO2, blood pressure, perceived fatigue, and respiratory function tests.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy between the ages of 18-25,
* Volunteering to participate in the study,
* Signing the voluntary consent form,
* Being an amateur football player who continues his/her active sports life,
* Not having an injury that prevents participation in the study.

Exclusion Criteria:

* Having a disease related to the respiratory system,
* Having a disease related to the cardiac system,
* Having any chronic disease and using a medication related to it.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Respiratory Function Test | 2 Months
  In our study, FVC measurement were calculated using a MiniSpir2 brand spirometer device. The measurements were performed while the participants were sitting in a fixed chair. The measurements were repeated 3 times for each participant and the two highest values read on the device were recorded as an average.
Respiratory Function Test | 2 Months
  In our study, FEV1/FVC measurement were calculated using a MiniSpir2 brand spirometer device. The measurements were performed while the participants were sitting in a fixed chair. The measurements were repeated 3 times for each participant and the two highest values read on the device were recorded as an average.
Respiratory Function Test | 2 Months
  In our study, PEF measurement were calculated using a MiniSpir2 brand spirometer device. The measurements were performed while the participants were sitting in a fixed chair. The measurements were repeated 3 times for each participant and the two highest values read on the device were recorded as an average.
Respiratory Function Test | 2 Months
  In our study, FEV1 measurement were calculated using a MiniSpir2 brand spirometer device. The measurements were performed while the participants were sitting in a fixed chair. The measurements were repeated 3 times for each participant and the two highest values read on the device were recorded as an average.

SECONDARY OUTCOMES:
BORG Perceived Fatigue Measurement | 2 Months
  The Borg Perceived Fatigue Scale was used to assess the degree of fatigue perceived by the participants. BORG is a scale developed to assess the level of strain experienced by individuals during physical activities. This scale is based on physical measures such as respiratory rate, heart rate, muscle fatigue and sweating perceived by individuals during physical exertion. The scale is scored between 6 and 20. If the participant's perceived muscle fatigue is very mild, a score of 9 is given. Scores between 12 and 14 on BORG indicate that the exertion is moderate. If the individual perceives that they are exerting very much, a score of 19 is given.

OTHER OUTCOMES:
Pulse Measurement | 2 Months
  Endostall Pulse Oximeter device was used to measure the participants' pulse values.
SPO2 Measurement | 2 Months
  Endostall Pulse Oximeter device was used to measure the participants' SPO2 values.
Blood Pressure Measurement | 2 Months
  Systolic and diastolic blood pressures of all participants were measured using an Omron M6 AC HEM-7322-E arm blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: ALİ KARAAĞAÇ, MSc, Principal Investigator — Principal Investigator
Locations (1):
- İstanbul Gelisim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No